CLINICAL TRIAL: NCT07182695
Title: Effect of Bilateral Cervical Erector Spinae Plane Block on Dyspnea in Patients With Acute Respiratory Failure: A Prospective Single-Cohort Study
Brief Title: Cervical Erector Spinae Plane Block for Dyspnea in Acute Respiratory Failure: A Prospective Cohort
Status: Not yet recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Çağrı Arslan, Principal Investigator, Hacettepe University
Other Study IDs: KA-25017
Record Dates: First submitted 2025-09-04; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Acute Respiratory Failure (ARF); Dyspnea
Keywords: Cervical ESP block; Diaphragm ultrasound; Intensive care; Ultrasound-guided regional anesthesia
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cervical ESP cohort: adults with acute respiratory failure receiving bilateral cervical ESP block

SUMMARY:
Dyspnea is common and distressing in patients with acute respiratory failure. In our intensive care unit, some patients receive a cervical erector spinae plane (ESP) block to help relieve dyspnea. This study will observe patients who receive bilateral cervical ESP blocks and measure changes in dyspnea using validated scales at predefined time points over 24 hours. We will also track vital signs, arterial blood gas values, and diaphragm movement on ultrasound.

DETAILED DESCRIPTION:
Prospective, single-cohort observational study in an adult ICU. Consecutive eligible patients with acute respiratory failure who receive bilateral cervical ESP block will be enrolled. Dyspnea severity will be measured using a 100-mm Dyspnea Visual Analog Scale (D-VAS), the Respiratory Distress Observation Scale (RDOS), and the Intensive Care RDOS (IC-RDOS) before the block (baseline) and at 30 minutes, 8 hours, 16 hours, and 24 hours after the block. Vital signs (respiratory rate, heart rate, peripheral oxygen saturation, blood pressure) will be recorded at the same time points. From arterial blood gases, pH, PaO₂, PaCO₂, SaO₂, and HCO₃- will be abstracted. Bilateral diaphragm excursion amplitude will be measured with bedside ultrasound. Statistical plan includes normality checks; repeated-measures ANOVA for parametric data or Friedman test for nonparametric data; paired t-test or Wilcoxon as needed; chi-square or Fisher's exact for categorical variables. Planned sample size: 30 (power analysis for repeated measures with effect size 0.25, α=0.05, power=0.90).

ELIGIBILITY:
Inclusion Criteria:

* ICU admission with acute respiratory failure.
* Patient or legally authorized representative provides consent.
* Cervical ESP block performed for dyspnea treatment

Exclusion Criteria:

* Infection at block site.
* Known diaphragm paralysis.
* Known allergy to local anesthetics.
* Refusal of consent (patient or representative).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients in the mixed medical-surgical ICU of a tertiary university hospital (Hacettepe University Hospital, Ankara, Türkiye). The ICU manages acute respiratory failure due to pneumonia, COPD/asthma, pulmonary edema, and post-operative causes. Patients who receive a cervical ESP block for dyspnea as are observed for changes over 24 hours.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Change in Dyspnea by Visual Analog Scale (D-VAS) | Baseline (pre-block), 30 minutes, 8 hours, 16 hours, and 24 hours after the ESP block.
  Patient-reported dyspnea on a 100-mm line (0=no dyspnea, 100=worst imaginable); measured in mm from 0 anchor to the patient's mark.

SECONDARY OUTCOMES:
Respiratory Distress Observation Scale (RDOS) Score | Baseline, 30 minutes, 8 hours, 16 hours, 24 hours post-block.
  Observer-rated RDOS (higher scores indicate more severe respiratory distress); standard scoring per instrument.
Intensive Care Respiratory Distress Observation Scale (IC-RDOS) Score | Baseline, 30 minutes, 8 hours, 16 hours, 24 hours post-block.
  Observer-rated IC-RDOS (higher scores worse); standard scoring per instrument.
Diaphragm Excursion Amplitude on Ultrasound | Baseline (pre-block), 30 minutes
  Peak-to-peak diaphragm excursion amplitude measured bilaterally with bedside ultrasound/M-mode.
Arterial Blood Gas Parameters: pH, PaO₂, PaCO₂ , SaO₂, HCO₃- | Baseline (pre-block), 30 minutes, 8 hours, 16 hours, and 24 hours after the ESP block.
  Abstracted from ABGs
Adverse Events Related to ESP Block | From block through 24 hours.
  Number of participants with any block-related AE within 24 hours, per chart review/clinical documentation.
Respiratory Rate (Breaths/minute) | Baseline, 30 minutes, 8 hours, 16 hours, 24 hours post-block.
  Respiratory Rate recorded per routine monitoring.
Heart Rate (Beats/minute) | Baseline, 30 minutes, 8 hours, 16 hours, 24 hours post-block.
  Heart rate recorded per routine monitoring.
SpO₂ (%) | Baseline, 30 minutes, 8 hours, 16 hours, 24 hours post-block.
  SpO₂ recorded per routine monitoring.
Blood Pressure (mm-Hg) | Baseline, 30 minutes, 8 hours, 16 hours, 24 hours post-block.
  Blood Pressure recorded per routine monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Seda Banu AKINCI, Professor, Principal Investigator — Hacettepe University

IPD SHARING:
Plan to Share IPD: Undecided